CLINICAL TRIAL: NCT01047618
Title: The Incidence and Risk Factors of Venous Thromboembolism in Advanced Gastric Cancer Patients: Prospective Observational Study
Brief Title: Venous Thromboembolism in Advanced Gastric Cancer Patients
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Other Study IDs: AMC0904
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Advanced Gastric Cancer
Keywords: venous thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thromboembolism

SUMMARY:
Venous thromboembolism (VTE), which includes pulmonary embolism (PE) and deep vein thrombosis (DVT), is a common complication and leading cause of death in cancer patients. Large, population-based studies have shown that patients with cancer have four- to seven-fold increased risk of developing VTE compared with patients without cancer. VTE would be frequent in patients with advanced gastric cancer, especially associated chemotherapy. However, relatively few studies have been conducted regarding the incidence of VTE in Asian cancer patients. According to previous review, Asian patients significantly lower risk of developing VTE. The rate of VTE with advanced gastric cancer, and associated chemotherapy is not known in Asian patients. In addition, the impact of VTE on overall survival has not been documented in these patients.

DETAILED DESCRIPTION:
Primary objectives - To evaluate the incidence of VTE in advanced gastric cancer with chemotherapy and to identify risk factors and biomarkers for VTE in this population

Secondary objectives

- To investigate the significant impact of VTE on overall survival and in this population

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented gastric adenocarcinoma including adenocarcinoma of the gastro-esophageal junction
* Age 18 years or older
* Locally advanced (inoperable) or metastatic gastric cancer, initially diagnosed, recurrent gastric cancer
* Performance status (ECOG scale) : 0-2
* Adequate bone marrow function:
* Adequate renal function
* Adequate hepatic function:
* Required to be at the start of a new chemotherapy regimen
* Received chemotherapy one cycle or more
* Adequate follow-up for at least 12 weeks
* Patients should sign a written informed consent before study entry

Exclusion Criteria:

* Previously exposed to chemotherapy exception adjuvant or neoadjuvant therapy
* Second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence
* Prior radiotherapy was administered to target lesions selected for this study, or radiotherapy to the non-target lesions has been completed within 4 weeks before randomization
* Presence of CNS metastasis
* Major surgery within 4 weeks before initiation of study treatment or lack of complete recovery from the effects of major surgery. Patient received curative operation or RFA for metastatic disease.
* Significant traumatic injury within 4 weeks prior to enrollment
* Serious illness or medical conditions, as follows:

  1. Congestive heart failure (NYHA class III or IV)
  2. Unstable angina or myocardial infarction within the past 12 months
  3. Significant arrhythmia requiring medication and conduction abnormality such as over 2nd degree AV block
  4. Uncontrolled hypertension
  5. Liver cirrhosis (≥ Child class B)
  6. Psychiatric disorder that may interfere with protocol compliance
  7. Unstable diabetes mellitus
  8. Active infection
* Superficial thrombophlebitis, transient ischemic attacks, and thrombosis occurring in setting of disseminated intravascular coagulation
* Pregnant or lactating women
* Hormonal replacement therapy within 4 weeks
* Chronic oral treatment with corticosteroid unless initiated > 6 months prior to study entry and at low dose (≤ 20mg methylprednisolone or equivalent)
* Warfarin of heparin therapy
* Not able or willing to give informed consent
* Any patients judged by the investigator to be unfit to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of advanced gastric cancer with palliative chemotherapy
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2009-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of VTE in advanced gastric cancer with chemotherapy and to identify risk factors and biomarkers for VTE in this population | 2 years

SECONDARY OUTCOMES:
To investigate the significant impact of VTE on overall survival and in this population | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Koo Kang, MD,PhD, Principal Investigator — Asan Medical Center; Baek-Yeol Ryoo, MD,PhD, Principal Investigator — Asan Medical Center; Min-Hee Ryu, MD,PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea